CLINICAL TRIAL: NCT05901454
Title: Yellow Fever Human Infection Model With YF-17D
Acronym: YF-INFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: The International Society of Travel Medicine (Unknown)
Responsible Party: Principal Investigator, Anna HE Roukens, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL70951.058.19
Record Dates: First submitted 2023-05-23; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Intervention Model Description: human infection model of yellow fever with the yellow fever 17D vaccine and viruria (virus in urine) as readout
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention arm (Other): yellow fever vaccine arm (all participants receive the standard yellow fever vaccine (Stamaril)
  Interventions: Drug: Yellow Fever Vaccine

INTERVENTIONS:
Drug: Yellow Fever Vaccine — vaccination according to manufacturers manual (0.5mL subcutaneously in the arm)
  Other Names: Stamaril (yellow fever vaccine)

SUMMARY:
No antiviral treatment exists for yellow fever, only supportive care, and therefore we rely on prevention through vaccination. Although this vaccine is very effective, stockpiles are insufficient in outbreak situations and some people have a contraindication to be vaccinated. For those who are unprotected and at risk of yellow fever infection, treatment could be life saving.

DETAILED DESCRIPTION:
No antiviral treatment exists for yellow fever, only supportive care, and therefore we rely on prevention through vaccination. Although this vaccine is very effective, stockpiles are insufficient in outbreak situations and some people have a contraindication to be vaccinated. For those who are unprotected and at risk of yellow fever infection, treatment could be life saving.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years

Exclusion Criteria:

* contraindication to receive YF-17D (immune deficiency, thymus illness)
* previous YF vaccination
* pregnancy
* chicken egg allergy
* hypersensitivity to any other substance in the YF-17D vaccine
* interval of < 4 weeks of another live attenuated vaccine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
yellow fever 17D in urine | within 30 days of the vaccination
  yellow fever 17D in urine at sequential time points after vaccination

SECONDARY OUTCOMES:
peak of YF 17D viruria after vaccination | within 30 days of the vaccination
  days after vaccination on which most participants have a positive yellow fever virus PCR on urine as material
YF-17D viremia (in plasma) after vaccination | within 14 days of the vaccination
  days after vaccination on which most participants have a positive yellow fever virus PCR on plasma as material

CONTACTS AND LOCATIONS:
Overall Officials: Anna HE Roukens, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
research protocol and data will be shared upon request according to the institution's (LUMC) policy